CLINICAL TRIAL: NCT01217905
Title: A Phase I, Single Centre, Single-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD7687 After Administration of Single and Multiple Ascending Doses in Healthy Male Japanese Subjects
Brief Title: Japanese Single and Multiple Ascending Dose, Safety, Tolerability, Pharmacokinetic (PK) & Pharmacodynamic (PD) Study of AZD7687
Acronym: JSMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: D2710C00004
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Phase 1; Type 2 diabetes; obesity; Japanese healthy volunteer; AZD7687
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — AZD7687

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD7687

INTERVENTIONS:
Drug: AZD7687 — Oral suspension

SUMMARY:
This is a study in Japanese healthy volunteers to determine the safety and tolerability of the compound AZD7687. It will also assess how the body handles the drug and how it responds to the drug following single dose followed by multiple dosing over 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between 19 and 35 kg/m2 and weigh at least 50 kg and no more than 90 kg
* Male subjects should be willing to use barrier contraception ie, condoms with spermicide, from the first day of dosing until 3 months after the last dose of investigational product

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational product

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Investigate the safety and tolerability of AZD7687 following administration of single and multiple doses | From screening period to follow-up visit 45 days (Maximum).

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics (PK) (plasma and urine) of AZD7687 and it´s glucuronic acid metabolite (AZ13128940) after single and multiple doses | Before dose and repeatedly to follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD MFPM FRCA, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Research site, Croydon, United Kingdom